CLINICAL TRIAL: NCT01635517
Title: Multicenter Tolvaptan Study For Uncontrolled Volume Overload in Japanese Acute Decompensated Heart faIlure Patients: A Prospective Observational Multicenter Cohort Study
Brief Title: Efficacy and Safety of Tolvaptan in Japanese Patients With Acute Heart Failure
Acronym: MT FUJI
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Nippon Medical School, Musashi Kosugi Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRIHF1203; UMIN000008258 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure
Keywords: Diuretics; Vasopressins; Sodium
MeSH Terms: conditions — Heart Failure; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tolvaptan: Tolvaptan administration

SUMMARY:
The aims of the present study are to investigate prospectively the clinical course and outcome of the hospitalized heart failure patients treated with tolvaptan for management of fluid retention and serum sodium levels of less than 140 mEq/L and also to analyze the factors related with the efficacy including outcome of tolvaptan therapy.

DETAILED DESCRIPTION:
Vasopressin mediates fluid retention in heart failure. Tolvaptan, an oral, nonpeptide, selective vasopressin V2-receptor antagonist, shows promise for management of heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. hospitalized patients for decompensated heart failure with signs of fluid retention despite using diuretics other than tolvaptan and planned tolvaptan use
2. serum Na < 140 mEq/L
3. age: > or = 20 years at the time of informed consent
4. provided written informed consent.

Exclusion Criteria:

1. hemodynamic instability
2. patients with hypersensitivity to tolvaptan or similar compounds
3. anuric patients
4. patients who cannot feel thirst and are difficult to intake the fluid
5. patients who are pregnant, potentially pregnant or willing to be pregnant
6. patients have taken tolvaptan before enrollment after hospitalization
7. acute coronary syndrome
8. adrenal insufficiency
9. patients scheduled to undergo coronary angioplasty within the study period
10. ineligible patients according to the investigator's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for decompensated heart failure with fluid retention and serum sodium levels of less than 140 mEq/L
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy 1) Alleviation of the signs of body fluid retention 2) Change of body weight 3) Changes in the daily urinary volume | At the day of discontinuation of tolvaptan or day 7, whichever comes first
  1) Alleviation of the signs of body fluid retention by the 7th day of treatment with tolvaptan (or the day of discontinuation of the drug in cases where tolvaptan treatment has been discontinued before the 7th day) as compared with the observations made on the day before the start of treatment 2) Change of body weight by the 7th day of treatment with tolvaptan as compared with the level measured on the day before the start of treatment 3) Changes in the daily urinary volume by the 7th day of treatment with tolvaptan as compared with the values measured on the day before the start of treatment
Safety: adverse events Adverse events until 30 days after the end of treatment with tolvaptan | 30 days after tolvaptan withdrawal
Long-term outcome (1 year after tolvaptan administration) 1) Time from enrollment to cardiovascular events 2) Time from enrollment to re-hospitalization for aggravation of heart failure 3) Time from enrollment to all-cause death | 1 year after administration of tolvaptan
  1) Time from enrollment to cardiovascular events within 1 year after administration of tolvaptan 2) Time from enrollment to re-hospitalization for aggravation of heart failure within 1 year after administration of tolvaptan 3) Time from enrollment to all-cause death within 1 year after administration of tolvaptan
  Cardiovascular events included death from heart failure, death from acute coronary syndrome, death from stroke, sudden death, death of unknown causes, death from other cardiovascular causes, readmission for heart failure, ventricular arrhythmia, acute coronary syndrome, and stroke.

SECONDARY OUTCOMES:
Search for the factors related with the efficacy of tolvaptan therapy and long-term outcome 1) related factors regarding efficacy of tolvaptan 2 ) related factors regarding long-term outcome | 1 year after administration of tolvaptan
  Exploratory analysis will be performed to determine which factors relate with the efficacy of tolvaptan therapy or long-term outcome. Factors will include age, gender, medical past history, medication, NYHA classification, Nohria/Steavenson classification, laboratory data (Na, K, Cl, Albumin, Cr, BUN, AST, ALT, gamma-GTP, LDH, T-Bil, BNP, NT-pro BNP, copeptin, galectin-3,aldosteron,angiotensin II, renin, noradrenaline), heart rate, blood pressure, echocardiography data, intake/urine volume and osmolality.

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Sato, MD,PhD, Principal Investigator — Nippon Medical School, Musashi Kosugi Hospital
Locations (1):
- Nippon Medical School, Musashi Kosugi Hospital, Kawasaki, Kanagawa, Japan